CLINICAL TRIAL: NCT05394922
Title: Glycosylation Analysis of Anti-DNA Auto-antibodies as Biomarker in the Follow up of Patients With Lupus Erythematosus Disseminated (GALA)
Brief Title: Glycosylation Analysis of Lupus Anti-DNA Antibodies (GALA)
Acronym: GALA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0404
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Lupus Erythematosus Disseminatus; Autoimmune Diseases; Chronic Disease
Keywords: lupus erythematosus; autoantibody; anti-dna antibody; glycosylation
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systemic lupus erythematosus (SLE) is a severe autoimmune disease in which patients often develop numerous autoantibodies (Abs). Unfortunately, none of the SLE specific Abs described so far (anti-DNA, -C1q, -nucleosome) are correlated enough to the disease activity to be used as a useful biomarker and reliably help in the therapeutic decision.

Abs effector functions, including antibody-dependent cell-mediated cytotoxicity (ADCC), antibody-dependent cellular phagocytosis (ADCP) and antibody-mediated complement activation, are conditioned by the structure of the crystallizable fragment (Fc) and especially the N-linked oligosaccharide structures attached to the asparagine-297 in the CH2 domain of the Fc region. It has been shown that the decrease in galactosylation, sialylation and fucolylation is generally associated with inflammatory function of circulating IgG whereas Abs with sialic acid, fucose and/or galactose in Asn-297 are anti-inflammatory. This major role of Ab glycosylation in the regulation of the effector and pathogenic functions of Abs have been well documented in rheumatoid arthritis and ANCA associated vasculitis with a good correlation between Ab sialylation and disease activity. In lupus, it has been shown that glycosylation of total IgG is also altered and correlated with disease activity but glycosylation analysis of the LES specific Abs is still lacking.

The aim of this study is to analyse by mass spectrometry (MS) the different glycoforms of anti-DNA Abs in lupus patients and find a correlation with disease activity.

DETAILED DESCRIPTION:
140 adult patients with lupus and anti-DNA Abs will be prospectively recruited in the University Hospital of Montpellier and Nîmes (department of rheumatology, internal medicine and nephrology) and followed during 1 year.

Blood samples will be drawn at inclusion, at 1 year and during any flare of the disease. After centrifugation (2000g x 10 minutes) serum will be aliquoted and frozen at -80°C.

At the end of the study, total IgG will be isolated using protein G and anti-DNA Abs will be purified from total IgG with DNA affinity columns. Glycosylation status of the anti-DNA Abs will be extensively determined by mass spectrometry and correlated to disease activity (SLEDAI).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with LED according to the ACR/EULAR 2019 criteria, all clinical forms combined, quiescent or in flare with positive native anti-DNA antibodies, providing oral informed consent.

Exclusion Criteria:

* Patients under protection of justice or unable to receive a clear information.
* High probability of non-compliance with the protocol or withdrawal during the study
* Already involved in another interventional clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting with LED according to the ACR/EULAR 2019 criteria, all clinical forms combined, quiescent or in flare with positive native anti-DNA antibodies, providing oral informed consent
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
anti-DNA glycoform measurement at inclusion | inclusion
  measurement of the serum concentration of the different anti-DNA Ab glycoforms at inclusion and correlation with disease activity

SECONDARY OUTCOMES:
anti-DNA glycoform measurement at 1 year | 1 year
  measurement of the serum concentration of the different anti-DNA Ab glycoforms after 1 year and correlation with disease activity
anti-DNA glycoform measurement during a flare | 1 year
  measurement of the serum concentration of the different anti-DNA Ab glycoforms during any flare of the disease and correlation with disease activity

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Montpellier University Hospital, Montpellier
  - Nimes University Hospital, Nîmes